CLINICAL TRIAL: NCT06745154
Title: QUEST (Quitting Using Executive Function Strategy Training) Research Protocol
Brief Title: Evaluating the Impact of Quitting Using Executive Function Strategy Training (QUEST) on Smoking Cessation in Homeless Young Adult Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OSU-23119; NCI-2024-04793 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Cigarette Smoking-Related Carcinoma
MeSH Terms: interventions — Specimen Handling; Mental Status and Dementia Tests; Interviews as Topic; Nicotine Replacement Therapy; Smoking Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prevention (QUEST) (Experimental): Patients receive access to the Ohio Tobacco Quitline, receive nicotine patches, gum, or lozenges for up to 8 weeks. Patients also participate in tobacco cessation counseling sessions for 5 sessions over 8 weeks. Patients additionally undergo cognitive assessment and nasal swab collection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Cognitive Assessment; Other: Interview; Drug: Nicotine Replacement; Behavioral: Smoking Cessation Intervention; Other: Survey Administration; Other: Tobacco Cessation Counseling

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo nasal swab collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Cognitive Assessment — Undergo cognitive assessment
Other: Interview — Ancillary studies
Drug: Nicotine Replacement — Given nicotine patches, gum, or lozenges
  Other Names: Nicotine Replacement Therapy; NRT
Behavioral: Smoking Cessation Intervention — Receive access to the Ohio Tobacco Quit Line
  Other Names: Smoking and Tobacco Use Cessation Interventions
Other: Survey Administration — Ancillary studies
Other: Tobacco Cessation Counseling — Participate in counseling sessions

SUMMARY:
This clinical trial evaluates the impact of Quitting Using Executive Function Strategy Training (QUEST) on quitting smoking (cessation) in homeless young adult smokers with an acquired brain injury (ABI). Over 70% of youth and young adults experiencing homelessness (YYEH) smoke tobacco. More than half of YYEH who smoke have made at least one attempt to quit smoking but few use evidence-based methods to increase success. In addition, 9 out of 10 of these have an acquired brain injury which may have a negative impact on successful smoking cessation. QUEST may help homeless young adult smokers with an ABI quit smoking.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Gather data needed to build QUEST (Quitting Using Executive function Strategy Training), an intervention to help youth and young adults (YYEH) with executive function dysregulation better 1) access evidence-based cessation; 2) adhere to processes of evidence-based treatment; and 3) address stress to prevent relapse.

II. Establish the feasibility of collecting acquired brain injury (ABI) status, and impact data sensitive to change over time (clinical and epigenetic), from YYEH tobacco users in community settings.

EXPLORATORY OBJECTIVE:

I. Determine if 1) executive functioning 2) mild cognitive impairment and 3) epigenetic age & other biomarkers of health risk measures are sensitive to difference by ABI status among YYEH past week combustible tobacco users.

OUTLINE:

Patients receive access to the Ohio Tobacco Quitline, receive nicotine patches, gum, or lozenges for up to 8 weeks. Patients also participate in tobacco cessation counseling sessions for 5 sessions over 8 weeks. Patients additionally undergo cognitive assessment and nasal swab collection on study.

ELIGIBILITY:
Inclusion Criteria:

* 18-24 years old
* Utilizing STAR House ( a drop-in center for youth and young adults experiencing homelessness) services
* Use of combustible tobacco product in the last week
* Willing to quit smoking in the next 30 days
* Acquired Brain Injury (ABI) (15 youth with and 15 without)

  * CHATS will be used to determine ABI. Ask "C", "H" and "A" of the CHATS tool. If yes to C OR H and yes to A, that will be considered positive for ABI
* Have access to a phone
* Willing to use phone for QuitLine (QL) services
* Willing to enroll in Ohio Tobacco Quit Line
* Willing to share Ohio Tobacco Quit Line portal data with researchers
* Willing to provide biospecimens (exhaled air and nasal samples)
* Conversational English skills

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Rate of executive function difficulties | Up to 8 weeks
  The number of times participants experience executive function difficulties with adhering to the Quit Line protocol will be recorded via survey questionnaires.
Factors impacting access to evidence-based treatment | Up to 8 weeks
  All factors reported by participants via survey questionnaires that impacted their ability to access Quit Line treatment will be recorded.
Contact with Quitline | Up to 8 weeks
  The number of contacts each participant had with the Quit Line throughout the study will be recorded via survey questionnaires.
Use of nicotine replacement therapy | Up to 8 weeks
  The number of times participants made use of nicotine replacement therapies throughout the length of the study will be recorded via survey questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Julianna Nemeth, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu